CLINICAL TRIAL: NCT03064165
Title: Postoperative Analgesia After Elective Hip Surgery - Effect of Obturator
Brief Title: Postoperative Analgesia After Elective Hip Surgery - Effect of Obturator Nerve Blockade
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Elective Surgery Centre, Silkeborg Regional Hospital (Unknown)
Responsible Party: Principal Investigator, Niels Dalsgaard Nielsen, MD, PhD-fellow, University of Aarhus
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HIP/FUSION#2
Record Dates: First submitted 2017-02-13; First posted 2017-02-24 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Obturator Nerve Block; Total Hip Replacement
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Obturator nerve block (Experimental): Postoperative obturator nerve block with 15 mL bupivacain 5 mg/mL and epinephrine 5 µg/mL.
  Interventions: Drug: Bupivacaine-epinephrine; Procedure: Obturator nerve block
- Sham block (Placebo Comparator): Postoperative sham-block with normal saline.
  Interventions: Procedure: Sham block; Drug: Sodium Chloride 9mg/mL

INTERVENTIONS:
Drug: Bupivacaine-epinephrine — Nerve block with 15 mL bupivacain 5 mg/mL with epinephrine 5 µg/mL.
  Arms: Obturator nerve block
Procedure: Sham block — Injection as for obturator nerve block, but with placebo
  Arms: Sham block
Procedure: Obturator nerve block — Postoperative obturator nerve block
  Arms: Obturator nerve block
Drug: Sodium Chloride 9mg/mL — Placebo
  Arms: Sham block

SUMMARY:
The study investigates the effect of an obturator nerve block on the postoperative pain and opioid consumption after total hip replacement.

ELIGIBILITY:
Inclusion Criteria:

* Patients for primary hip replacement in spinal anesthesia
* Age >= 18 years
* American Society of Anesthesiologists physical status classification score I-III
* Informed consent

Exclusion Criteria:

* Lacking the ability to corporate
* Lacking the ability to speak danish
* Planned discharge on the same day of surgery
* Neuropathy of the lower extremities
* Contraindications for NonSteroidal Anti-Inflammatory Drugs (NSAID)
* Contraindications for dexamethasone
* Chronic opioid demanding pain
* Pregnancy
* Allergy towards one or both investigatory medicinal products
* Active treatment with amiodarone
* Active treatment with verapamil
* Active treatment with corticosteroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2018-06-08 (Actual); Study Completion 2018-06-08 (Actual)

PRIMARY OUTCOMES:
Opioid dose 0-12 hour after total hip replacement | 0-12 hour after completion of total hip replacement
  Cumulated dose of opioid 0-12 hour after total hip replacement

SECONDARY OUTCOMES:
Cumulated dose of opioid 12-18 hours after total hip replacement. | 12-18 hours after completion of total hip replacement
Pain at rest at time of examination (numeric rating scale) | 1, 2, 5, 7 and 24 hours after completion of total hip replacement
Pain at passive 90-degree hip flexion (numeric rating scale) | 1, 2, 5, 7 and 24 hours after completion of total hip replacement
Worst pain during ambulation on the day of surgery | 5 hours after completion of total hip replacement
Time from completion of surgery to first dose of opioid | 24 hours after completion of total hip replacement
Intensity of nausea on time of examination (numeric rating scale) | 1, 2, 5, 7 and 24 hours after completion of total hip replacement
Incidences of emesis 0-18 hours after total hip replacement. | 0-18 hours after completion of total hip replacement
Cumulated dose of ondansetron 0-18 hours after total hip replacement | 0-18 hours after completion of total hip replacement
Cumulated dose of droperidol 0-18 hours after total hip replacement | 0-18 hours after completion of total hip replacement
Length of stay on post anesthesia care unit after completion of total hip replacement | 24 hours after completion of total hip replacement
Length of stay on hospital after completion of total hip replacement | Up to 2 days
Ability to ambulate 5 hours after surgery | 5 hours after completion of total hip replacement
  Ability to sit, stand, walk with tall rollator and walk with crutches
Motor control with operated leg | 5 hours after completion of total hip replacement
  Physiotherapist evaluating motor control with operated leg during ambulation.
Self-reported sleep quality the first night after total hip replacement | 24 hours after completion of total hip replacement
  Self-reported sleep quality on a 3-point-scale: 2 = Undisturbed sleep; 1 = Sleep disturbed by other reasons than pain; 0 = Sleep disturbed by pain.
Duration of spinal anesthesia | 0-4 hours after completion of total hip replacement
  Time from end of operation until regain of normal sensibility on anterior femur.

CONTACTS AND LOCATIONS:
Locations (1):
- Elective Surgery Centre, Silkeborg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared through the Danish Data Archive.

REFERENCES:
- [Derived] Nielsen ND, Runge C, Clemmesen L, Borglum J, Mikkelsen LR, Larsen JR, Nielsen TD, Soballe K, Bendtsen TF. An Obturator Nerve Block does not Alleviate Postoperative Pain after Total Hip Arthroplasty: a Randomized Clinical Trial. Reg Anesth Pain Med. 2019 Jan 23:rapm-2018-100104. doi: 10.1136/rapm-2018-100104. Online ahead of print. PMID 30679337